CLINICAL TRIAL: NCT03564730
Title: Randomized Control Trial of Staged Versus Simultaneous Bilateral Total Knee Arthroplasty
Brief Title: Staged Versus Simultaneous Bilateral Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Innovation Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-046
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
Keywords: Bilateral, staged, simultaneous
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either simultaneous or staged bilateral KA procedures using randomly generated numbers permuted in blocks of 10.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Knee Arthroplasty (TKA) (Active Comparator): Patient will have complete replacement - Simultaneous vs Staged
  Interventions: Procedure: Simultaneous Knee Arthroplasty (UKA); Procedure: Staged Knee Arthroplasty (UKA)
- Unicompartmental Knee Arthroplasty (UKA) (Active Comparator): Patient will have half-knee replacement (partial) - Simultaneous vs Staged
  Interventions: Procedure: Simultaneous Knee Arthroplasty (UKA); Procedure: Staged Knee Arthroplasty (UKA)

INTERVENTIONS:
Procedure: Simultaneous Knee Arthroplasty (UKA) — Patient will have both knees completed under one anesthetic.
Procedure: Staged Knee Arthroplasty (UKA) — Patient will have knees completed under 2 anesthetics.

SUMMARY:
The purpose of this study is to assist surgeons and patients in answering the question "Should I have both knees replaced at the same time, or should I just do one and wait to do the second one?"

DETAILED DESCRIPTION:
This is a multi-center randomized controlled trial of 224 patients in order to clearly delineate differences in post-operative outcomes and the trajectory of recovery between simultaneous and staged bilateral KA. The primary outcome measure is difference in generic health related quality of life between the two groups measured 1 year following surgery. Secondary outcome measures include differences in joint specific scores, time off work, satisfaction and costs.

This trial will inform patients and clinicians about differences in recovery, function and efficacy of the procedure to aid in the selection of treatment pathway to best suit the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients considering bilateral knee arthroplasty
* Patients must sign the consent form
* Patients must be willing to complete the study questionnaires for the duration of the study

Exclusion Criteria:

* Patients who require simultaneous bilateral knee replacement surgery in order to manage significant bilateral flexion or valgus knee contractures where staged procedures may result in suboptimal outcomes by increasing the risk of post-operative flexion contracture in the "first replaced" knee
* patients who are unable to complete the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Veterans Rand 12-item Health Survey Score (VR-12) | 1 Year
  The VR-12 is a 12-item questionnaire corresponding to eight principal physical and mental health domains including general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy-fatigue, social functioning and mental health; patient-reported.

SECONDARY OUTCOMES:
Joint function (Oxford-12 knee score) | Pre-operative, 6 months, 12 months, 18 months, 24 months
  The Oxford Knee Score (OKS) is a patient self-administered 12-item questionnaire with each question having a Likaert-like response option (0-4). A total of the 12 items will indicated the joint function; lower total score = poorer function.
Return to work | Pre-operative, 6 months, 12 months, 18 months, 24 months
  Assessment of ability to return to work and time away from work following surgery.
Patient satisfaction | 6 months, 12 months, 18 months, 24 months
  Evaluate change in patient-reported satisfaction using a Likaert scale; 1=Very Satisfied to 5=Very Unsatisfied.
Complications | Intraoperative, 6 months, 12 months, 18 months, 24 months
  Evaluation type and frequency of complication (adverse events).
Hospital stay | Up to 1 week
  Number of days in hospital
Transfusion rate | Up to 1 week
  Number of unit transfused during hospital stay.
Costs of knee replacement surgery | Up to 1 week
  An attempt to calculate costs of surgery using length of stay data to calculate cost between Simultaneous vs Staged procedures. Length of stay will be calculated in days/hours.

CONTACTS AND LOCATIONS:
Overall Officials: Eric R. Bohm, MD, Principal Investigator — University of Manitoba
Locations (8):
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - Concordia Hospital, Winnipeg, Manitoba
  - St. Joseph's - McMaster University, Hamilton, Ontario
  - Kingston Health Sciences Center - KGH, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec